CLINICAL TRIAL: NCT03188380
Title: The Use of Different Imaging Modalities in Diagnosing Necrotizing Enterocolitis in Preterm Infants.
Brief Title: Imaging Modalities in Diagnosing Necrotizing Enterocolitis in Preterm Infants.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Princess Anna Mazowiecka Hospital, Warsaw, Poland (Other)
Collaborators: Jagiellonian University (Other); Ujastek Obstetrics and Gynaecology Hospital (Unknown); University Children's Hospital of Cracow (Unknown)
Responsible Party: Principal Investigator, Renata Bokiniec, Renata Bokiniec MD PhD, Princess Anna Mazowiecka Hospital, Warsaw, Poland
Other Study IDs: KAROWA USG VERSION 1.0
Record Dates: First submitted 2017-05-11; First posted 2017-06-15 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Necrotising Enterocolitis
Keywords: nec; abdominal ultrasound; abdominal radiograph; preterm
MeSH Terms: conditions — Enterocolitis, Necrotizing; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Plain abdominal radiograph (AR): After meeting enrolment criteria each patient will have an AR performed. One image will be obtained with a vertical beam and a horizontal beam, with the patient supine.
  Interventions: Diagnostic Test: Plain abdominal radiography; Diagnostic Test: Abdominal ultrasound
- Abdominal ultrasound (AUS): If plain abdominal radiography is inconclusive or no abnormalities typical for NEC are recorded, an AUS will be ordered.
  Interventions: Diagnostic Test: Plain abdominal radiography; Diagnostic Test: Abdominal ultrasound

INTERVENTIONS:
Diagnostic Test: Plain abdominal radiography — After meeting enrolment criteria each patient will have an AR performed. One image will be obtained with a vertical beam and a horizontal beam, with the patient supine.
Diagnostic Test: Abdominal ultrasound — If the AR is inconclusive or no abnormalities typical for NEC are recorded, an AUS will be ordered.

SUMMARY:
Background Necrotizing enterocolitis (NEC) is one of the most serious conditions in newborns, affecting up to 10% of very low birth weight infants (VLBW). In the most premature population mortality rates can rise as high as 60%.

Typical findings on abdominal radiography (AR) include pnuematosis intestinalis (PI), portal vein gas (PVG) and pneumoperitoneum, but are sometimes not present even in severe cases. Abdominal ultrasound (AUS) can depict PI, PVG and pnuemoperitoneum (in some cases a head of AR), but it also provides other crucial information such as bowel wall viability (thickness or thinning) and free abdominal fluid. These additional findings are helpful in expediting diagnosis and management of NEC.

Methods and analysis The hypothesis being tested is that preforming an AUR in patients with clinical symptoms of NEC but inconclusive/normal AR will enhance detection rates, and expedite treatment in infants born at <32 weeks.

Discussion The use of AUS together with AR as an add-on test may increase the accuracy of diagnosing NEC, and precipitate treatment. Swift implementation of antibiotics and bowel rest is extremely important. To our best knowledge, our study will be the first to focus only on VLBW, who are most prone to NEC. It will also be the first multi-centre study evaluating the use of AUS as an add-on test, enabling us to recruit a significantly higher number of patients compared to published studies.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal distension
* Visible bowels loops
* Feeding intolerance (defined as emesis ≥ 2 consecutive feeds, or gastric residuals of >50% per feed in ≥ 2 consecutive feeds, bilious residuals, bilious emesis)
* Temperature instability (defined as ≥ 2 consecutive measurements)
* Frank bloody stools
* Cardiovascular instability (hypotension; defined as MAP < 30mmHg, tachycardia >160/' or bradycardia < 80/')
* Recurrent apnea
* Increase of abdominal girth > 2cm (allowing inter-observer variability of 1 cm) within 12 h
* Abdominal wall erythemia

And/or at least 2 of the below laboratory findings5:

* Thrombocytopenia < 50 x103/uL
* Leukopenia <6 x106/uL
* CRP > 10 mg/L
* PCT > 1 ng/ml
* Coagulopathy

Exclusion Criteria:

* • < 22 weeks of gestational age or > 32 weeks (estimated by ultrasound)

  * Congenital abnormalities
  * No parental consent

Ages: 22 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: In this single-gate study we plan to include all consecutive preterm infants (born at <32 weeks of gestation) with suspected necrotizing enterocolitis based on the presence of at least three of the above mentioned clinical symptoms 4-7:
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Intervention time | until 40 weeks of post-conceptional age
  The time required to initiate conservative and/or surgical treatment after diagnosing NEC with AR versus AR and AUS

SECONDARY OUTCOMES:
Sensitivity and specificity | until 40 weeks of post-conceptual age
  Sensitivity and specificity of a diagnostic strategy involving a combination of AR (reference test) followed by AUS (index test) as compared to AR (reference test) in diagnosing NEC.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neonatology and Neonatal Intensive Care Warsaw Medical University, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided
All de-identified data collected during the trial will be available. The study protocol will also be available. These documents will be accessible to anyone who provides a methodologically sound proposal immediately following publication with no end date.

REFERENCES:
- [Derived] Seliga-Siwecka J, Rutkowski J, Margas W, Puskarz-Gasowska J, Bokiniec R. Sensitivity and specificity of different imaging modalities in diagnosing necrotising enterocolitis in a Polish population of preterm infants: a diagnostic test accuracy study protocol. BMJ Open. 2020 Jul 20;10(7):e033519. doi: 10.1136/bmjopen-2019-033519. PMID 32690727